CLINICAL TRIAL: NCT00271999
Title: Frequent Hemodialysis Network: Nocturnal Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Paul Eggers, Ph.D., Project Officer, NIH/NIDDK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: beck-night; 5U01DK066597 (NIH)
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: randomized controlled clinical trial; hemodialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Three times a week conventional at home hemodialysis
  Interventions: Behavioral: Nocturnal home hemodialysis
- 2 (Experimental): Six times a week nocturnal home hemodialysis
  Interventions: Behavioral: Nocturnal home hemodialysis

INTERVENTIONS:
Behavioral: Nocturnal home hemodialysis — Six times per week nocturnal home hemodialysis

SUMMARY:
The Frequent Hemodialysis (FHN) Nocturnal Trial is a randomized controlled trial recruiting subjects from dialysis units associated with designated Clinical Centers in the U.S. and Canada and followed for 12 months. Subjects will be randomized to conventional hemodialysis delivered three days per week home arm or to the six times per week nocturnal home hemodialysis arm which will follow any dialysis prescription provided their prescribed standardized Kt/V is at least 4.0 and treatment time is at least 6.0 hours, six times per week.

DETAILED DESCRIPTION:
This trial is a randomized, unblinded study of six times per week nocturnal home hemodialysis versus three times per week home hemodialysis. A target of 150 patients will be enrolled into this study with equal allocation in each arm, stratified by Clinical Center and residual renal function. All patients will be assessed for suitability for nocturnal home hemodialysis using a standardized method prior to patients entering the baseline portion of this protocol. The minimum dialysis dose in the standard arm will be an equilibrated Kt/V of 1.1 (equivalent to a standardized Kt/V (sKt/V) of 2.0) AND a minimum time of 2.5 hours. In the nocturnal arm there will be a minimum prescription of six hours per session for six days per week AND a minimum standardized Kt/V of 4.0. Patients will be followed for 12 months.

Two co-primary outcomes are designated: 1) a composite of mortality with the change over 12 months in the SF-36 RAND physical health composite, and 2) the change over 12 months in left ventricular mass. In addition, first priority secondary outcomes have been designated for seven outcome domains: 1) cardiovascular structure and function (change in LV mass), 2) physical function (change in the PHC), 3) depression/burden of illness (change in Beck Depression Inventory), 4) nutrition (change in serum albumin), 5) cognitive function (change in the Trail Making Test B), 6) mineral metabolism (change in average predialysis serum phosphorus), and 7) clinical events (rate of non-access hospitalization or death). Hypertension and anemia are also main outcome domains, but without designation of single first priority outcomes. The cost-effectiveness of the two interventions will also be compared.

The objectives of the study are as follows:

Feasibility:

1. To determine the feasibility of recruiting and retaining patients in a randomized trial of six times per week at-home nocturnal hemodialysis versus standard three times per week at home hemodialysis.
2. To determine patient adherence and acceptance of nocturnal hemodialysis, and to identify reasons for discontinuation or noncompliance to the interventions.

   Safety:
3. To determine the safety of the nocturnal hemodialysis intervention, with a particular emphasis on vascular access and patient burden.

   Efficacy:
4. To evaluate the efficacy of six times per week nocturnal HD compared to conventional three times per week HD on two co-primary outcomes: i) a composite of mortality with the change over 14 months in left ventricular mass by magnetic resonance imaging, and ii) a composite of mortality with the change over 14 months in the SF-36 RAND physical health composite score (PHC).
5. To determine the effect of six times per week nocturnal HD on nine secondary outcome domains: i) cardiovascular structure and function, ii) physical function, iii) depression/burden of illness, iv) nutrition, v) cognitive function, vi) mineral metabolism, vii) clinical events, viii) hypertension, and ix) anemia.

   Characterization of Interventions:
6. To characterize the six times per week nocturnal home hemodialysis intervention in comparison to standard home three times per week hemodialysis, including evaluation of small and middle molecule solute clearance, treatment time, and volume removal.

   Implementation:
7. To determine the feasibility of implementing six times per week nocturnal home hemodialysis in practice, including evaluation of barriers to implementation such as the home environment and any potential incremental costs of nocturnal home hemodialysis compared to three times per week conventional hemodialysis. An evaluation of the cost effectiveness of six times per week home nocturnal HD relative compared to 3 times per week conventional home HD will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end stage renal disease requiring chronic renal replacement therapy
2. Age ≥ 18 years,
3. Achieved mean eKt/V of ≥ 1.1 during Baseline

Exclusion Criteria:

1. GFR greater than 10 ml/min/1.73 m2 as measured by the average of urea and creatinine clearances obtained from a urine collection of at least 24 hours
2. Expectation that native kidneys will recover kidney function
3. Current access is temporary non-tunneled catheter
4. Unable to follow the nocturnal home hemodialysis training protocol for any reason, including inability to train the patient or the patient's caregiver
5. Non-compliance with hemodialysis or peritoneal dialysis treatments in the past
6. Medical conditions that would prevent the patient from performing the cardiac MRI procedure (e.g., inability to remain still for the procedure, a metallic object in the body, including cardiac pacemaker, inner ear (cochlear) implant, brain aneurysm clips, mechanical heart valves, recently placed artificial joints, and older vascular stents)
7. Unable to verbally communicate in English or Spanish
8. Current requirement for hemodialysis more than three times per week due to medical comorbidity (ultrafiltration session on fourth day per week not an exclusion criteria)
9. Currently on daily or nocturnal HD, or less than 3 months since the patient discontinued daily or nocturnal HD
10. Scheduled for living donor kidney transplant, change to peritoneal dialysis, or plans to relocate to an area outside of the referral area of one of the Clinical Centers within the next 12 months
11. Expected geographic unavailability at the Clinical Center (for standard arm patients) or at home (for nocturnal arm patients) for > 2 consecutive weeks or > 5 weeks total during the next 12 months (excluding unavailability due to hospitalizations)
12. Less than 3 months since the patient returned after acute rejection resulting in allograft failure
13. Currently in acute care or chronic care hospital
14. Life expectancy less than six months
15. A medical history that might limit the individual's ability to take trial treatments for the 12 month duration of the study, including: currently receiving chemo or radiotherapy for a malignant neoplastic disease other than localized non-melanoma skin cancer, active systemic infection (including tuberculosis, disseminated fungal infection, active AIDS but not HIV), and cirrhosis with encephalopathy
16. Current pregnancy or planning to become pregnant within the next fourteen months (patients require a higher dose of dialysis if pregnant). All female patients that have not gone through menopause will need to use an effective contraceptive method while enrolled in the study.
17. Contraindication to heparin, including allergy or heparin induced thrombocytopenia
18. Current use of investigational drugs or participation in an interventional clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial
19. Unable or unwilling to follow the study protocol for any reason (including mental incompetence)
20. Unable or unwilling to provide informed consent or sign IRB-approved consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
composite of 12 month mortality and the change over 12 months in left ventricular mass by cine-MRI, | 12 months
a composite of 12 month mortality and the change over 12 months in the SF-36 RAND physical health composite | 12 months

SECONDARY OUTCOMES:
cardiovascular structure/funct (change in LV mass over 12 mos), health-related QoL/phys funct (change over 12 mos in PHC), | 12 months
depression/dis burden (change over 12 mos in Beck Depression Inv.),nutrition (change over 12 mos in serum albumin, cognitive funct (change over 12 mos in TrailMaking Test B),mineral metabolism (change over 12 mos in aveg pre-dialysis serum phosphorus), | 12 months
clin events (rate of non-access hospital or death | 12 months
hypertension,anemia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. Eggers, Ph.D., Study Director — NIDDK, NIH; Michael V. Rocco, M.D., Principal Investigator — Wake Forest University; Gerald J. Beck, Ph.D., Principal Investigator — The Cleveland Clinic; Alan S. Kliger, M.D., Study Chair — Hospital of St. Raphael
Locations (1):
- Wake Forest University - Core center plus other centers in U.S. and Canada, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Suri RS, Garg AX, Chertow GM, Levin NW, Rocco MV, Greene T, Beck GJ, Gassman JJ, Eggers PW, Star RA, Ornt DB, Kliger AS; Frequent Hemodialysis Network Trial Group. Frequent Hemodialysis Network (FHN) randomized trials: study design. Kidney Int. 2007 Feb;71(4):349-59. doi: 10.1038/sj.ki.5002032. Epub 2006 Dec 13. PMID 17164834
- [Background] Kliger AS; Frequent Hemodialysis Network Study Group. High-frequency hemodialysis: rationale for randomized clinical trials. Clin J Am Soc Nephrol. 2007 Mar;2(2):390-2. doi: 10.2215/CJN.03110906. Epub 2006 Dec 20. No abstract available. PMID 17699439
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Chan CT, Kaysen GA, Beck GJ, Li M, Lo JC, Rocco MV, Kliger AS; FHN Trials. The effect of frequent hemodialysis on matrix metalloproteinases, their tissue inhibitors, and FGF23: Implications for blood pressure and left ventricular mass modification in the Frequent Hemodialysis Network trials. Hemodial Int. 2020 Apr;24(2):162-174. doi: 10.1111/hdi.12807. Epub 2019 Dec 11. PMID 31826326
- [Derived] Chan CT, Kaysen GA, Beck GJ, Li M, Lo J, Rocco MV, Kliger AS; FHN Trials. Changes in Biomarker Profile and Left Ventricular Hypertrophy Regression: Results from the Frequent Hemodialysis Network Trials. Am J Nephrol. 2018;47(3):208-217. doi: 10.1159/000488003. Epub 2018 Apr 5. PMID 29621747
- [Derived] Lo JC, Beck GJ, Kaysen GA, Chan CT, Kliger AS, Rocco MV, Li M, Chertow GM; FHN Study. Thyroid function in end stage renal disease and effects of frequent hemodialysis. Hemodial Int. 2017 Oct;21(4):534-541. doi: 10.1111/hdi.12527. Epub 2017 Mar 16. PMID 28301073
- [Derived] Garg AX, Suri RS, Eggers P, Finkelstein FO, Greene T, Kimmel PL, Kliger AS, Larive B, Lindsay RM, Pierratos A, Unruh M, Chertow GM; Frequent Hemodialysis Network Trial Investigators. Patients receiving frequent hemodialysis have better health-related quality of life compared to patients receiving conventional hemodialysis. Kidney Int. 2017 Mar;91(3):746-754. doi: 10.1016/j.kint.2016.10.033. Epub 2017 Jan 13. PMID 28094031
- [Derived] Lo JC, Beck GJ, Kaysen GA, Chan CT, Kliger AS, Rocco MV, Chertow GM; FHN Study. Hyperprolactinemia in end-stage renal disease and effects of frequent hemodialysis. Hemodial Int. 2017 Apr;21(2):190-196. doi: 10.1111/hdi.12489. Epub 2016 Oct 23. PMID 27774730
- [Derived] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Yang PC, Rajagopalan S; Frequent Hemodialysis Network Trial Group. Effects of frequent hemodialysis on ventricular volumes and left ventricular remodeling. Clin J Am Soc Nephrol. 2013 Dec;8(12):2106-16. doi: 10.2215/CJN.03280313. Epub 2013 Aug 22. PMID 23970131
- [Derived] Unruh ML, Larive B, Chertow GM, Eggers PW, Garg AX, Gassman J, Tarallo M, Finkelstein FO, Kimmel PL; FHN Trials Group. Effects of 6-times-weekly versus 3-times-weekly hemodialysis on depressive symptoms and self-reported mental health: Frequent Hemodialysis Network (FHN) Trials. Am J Kidney Dis. 2013 May;61(5):748-58. doi: 10.1053/j.ajkd.2012.11.047. Epub 2013 Jan 15. PMID 23332990
- [Derived] Kurella Tamura M, Unruh ML, Nissenson AR, Larive B, Eggers PW, Gassman J, Mehta RL, Kliger AS, Stokes JB; Frequent Hemodialysis Network (FHN) Trial Group. Effect of more frequent hemodialysis on cognitive function in the frequent hemodialysis network trials. Am J Kidney Dis. 2013 Feb;61(2):228-37. doi: 10.1053/j.ajkd.2012.09.009. Epub 2012 Nov 11. PMID 23149295
- [Derived] Hall YN, Larive B, Painter P, Kaysen GA, Lindsay RM, Nissenson AR, Unruh ML, Rocco MV, Chertow GM; Frequent Hemodialysis Network Trial Group. Effects of six versus three times per week hemodialysis on physical performance, health, and functioning: Frequent Hemodialysis Network (FHN) randomized trials. Clin J Am Soc Nephrol. 2012 May;7(5):782-94. doi: 10.2215/CJN.10601011. Epub 2012 Mar 15. PMID 22422538
- [Derived] Rocco MV, Lockridge RS Jr, Beck GJ, Eggers PW, Gassman JJ, Greene T, Larive B, Chan CT, Chertow GM, Copland M, Hoy CD, Lindsay RM, Levin NW, Ornt DB, Pierratos A, Pipkin MF, Rajagopalan S, Stokes JB, Unruh ML, Star RA, Kliger AS; Frequent Hemodialysis Network (FHN) Trial Group; Kliger A, Eggers P, Briggs J, Hostetter T, Narva A, Star R, Augustine B, Mohr P, Beck G, Fu Z, Gassman J, Greene T, Daugirdas J, Hunsicker L, Larive B, Li M, Mackrell J, Wiggins K, Sherer S, Weiss B, Rajagopalan S, Sanz J, Dellagrottaglie S, Kariisa M, Tran T, West J, Unruh M, Keene R, Schlarb J, Chan C, McGrath-Chong M, Frome R, Higgins H, Ke S, Mandaci O, Owens C, Snell C, Eknoyan G, Appel L, Cheung A, Derse A, Kramer C, Geller N, Grimm R, Henderson L, Prichard S, Roecker E, Rocco M, Miller B, Riley J, Schuessler R, Lockridge R, Pipkin M, Peterson C, Hoy C, Fensterer A, Steigerwald D, Stokes J, Somers D, Hilkin A, Lilli K, Wallace W, Franzwa B, Waterman E, Chan C, McGrath-Chong M, Copland M, Levin A, Sioson L, Cabezon E, Kwan S, Roger D, Lindsay R, Suri R, Champagne J, Bullas R, Garg A, Mazzorato A, Spanner E, Rocco M, Burkart J, Moossavi S, Mauck V, Kaufman T, Pierratos A, Chan W, Regozo K, Kwok S. The effects of frequent nocturnal home hemodialysis: the Frequent Hemodialysis Network Nocturnal Trial. Kidney Int. 2011 Nov;80(10):1080-91. doi: 10.1038/ki.2011.213. Epub 2011 Jul 20. PMID 21775973
- [Derived] Greene T, Daugirdas JT, Depner TA, Gotch F, Kuhlman M; Frequent Hemodialysis Network Study Group; National Institute of Diabetes and Digestive and Kidney Diseases; National Institutes of Health. Solute clearances and fluid removal in the frequent hemodialysis network trials. Am J Kidney Dis. 2009 May;53(5):835-44. doi: 10.1053/j.ajkd.2008.12.039. Epub 2009 Apr 1. PMID 19339093